CLINICAL TRIAL: NCT03778359
Title: Comparison of the Operation and Medical Treatment of Endometriosis and Adenomyosis
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-10-012AC
Record Dates: First submitted 2018-12-07; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Endometriosis; Adenomyosis
MeSH Terms: conditions — Endometriosis; Adenomyosis | interventions — Leuprolide; dienogest; Progestins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Gonadotropin-releasing hormone agonist treatment: Endometriosis post-operative Gonadotropin-releasing hormone agonist treatment
  Interventions: Drug: Leuprorelin
- Intrauterine device treatment: Endometriosis post-operative intrauterine device treatment
  Interventions: Device: Levonorgestrel
- Hormone therapy: Endometriosis post-operative hormone therapy
  Interventions: Drug: Dienogest
- Oral contraceptive: Endometriosis post-operative oral contraceptive
  Interventions: Drug: Progestins

INTERVENTIONS:
Drug: Leuprorelin — This study was designed to analyze the differences in prognosis and recurrence of patients with endometriosis and adenomyosis after receiving various surgical and medical treatments. This arm intervention is Leuprorelin.
  Groups: Gonadotropin-releasing hormone agonist treatment
Device: Levonorgestrel — This study was designed to analyze the differences in prognosis and recurrence of patients with endometriosis and adenomyosis after receiving various surgical and medical treatments. This arm intervention is Levonorgestrel.
  Groups: Intrauterine device treatment
Drug: Dienogest — This study was designed to analyze the differences in prognosis and recurrence of patients with endometriosis and adenomyosis after receiving various surgical and medical treatments. This arm intervention is Dienogest.
  Groups: Hormone therapy
Drug: Progestins — This study was designed to analyze the differences in prognosis and recurrence of patients with endometriosis and adenomyosis after receiving various surgical and medical treatments. This arm intervention is Progestins.
  Groups: Oral contraceptive

SUMMARY:
Endometriosis (including adenomyosis) is one of the most common gynecological diseases among women of childbearing age. Common symptoms such as menstrual pain, excessive menstrual flow, infertility, chronic lower abdominal pain, and painful intercourse. According to the literature statistics, the prevalence of endometriosis in women of childbearing age is about 10-20%, while the prevalence of adenomyosis is about 5%. Traditional medical treatments include hormones (danazol, gestrinone, oral lutein). Oral contraceptive, there is a Gonadotropin-releasing hormone agonist in the injection form, and a levonorgestrel-releasing intrauterine system in the intrauterine administration system. The choice of drugs has many influencing factors, such as the severity of endometriosis in patients (according to the classification of the American Society for Reproductive Medicine), the need for fertility, the convenience of drug use, and the patient's tolerance to drug side effects. Surgery is also one of the treatment options for endometriosis and adenomyosis, including traditional open or minimally invasive endoscopic ovarian cyst resection, oophorectomy, and lesion resection; adenomyosis surgery includes traditional methods Open abdominal, transvaginal or minimally invasive endoscopic hysterectomy, conservative uterine sparing adenomyomectomy and cytoreduction surgery (partial adenomyomectomy). For endometriosis, the common treatment consensus of obstetricians and gynecologists is to follow the surgical treatment of the lesions and then follow-up medication. For women with adenomyosis, if they have completed the birth, it is recommended to have a total hysterectomy, so that there is no recurrence. The possibility. However, for women who have not completed birth, conservative uterine preservation surgery is performed. According to research statistics, endometriosis or adenomyosis does not receive follow-up medical treatment after completion of surgical treatment, there is a high probability of recurrence, but the side effects caused by drugs will also affect the patient's compliance with medication.The Department of Women's Medicine of the hospital has a wealth of experience in the treatment of endometriosis and adenomyosis. Each year, about 500 cases of endometriosis (including adenomyosis) are performed. This study was designed to analyze the differences in prognosis and recurrence of patients with endometriosis and adenomyosis after receiving various surgical and medical treatments.

DETAILED DESCRIPTION:
The main purpose: to analyze the prognosis and treatment effect of endometriosis and adenomyosis after surgery and drug treatment.

Secondary objective: Analysis of endometriosis and adenomyosis after surgery and medication, the patient's assessment of drug side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endometriosis or adenomyosis-related surgery in the investigator's hospital from 2005/01/01 to 2018/12/31, and received follow-up medication.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects were patients who underwent endometriosis and adenomyosis-related surgery at Taipei Veterans General Hospital from 2005 to 2018. Review the surgical records and related medical records and record the follow-up medications received by the patients. The procedure includes traditional open or endoscopic ovarian cyst resection, oophorectomy, and lesion resection; open abdominal, transvaginal or endoscopic assisted transvaginal hysterectomy, open or endoscopic adenoma, gland Myomectomy. Postoperative patients received medication such as GnRH agonist, Levonorgestrel-releasing intrauterine system (LNG-IUS), hormonal preparation (danazol, gestrinone, oral lutein), oral Oral contraceptive, and tracking the size of the lesion with ultrasound, analyzing the patient's clinical prognosis, pain, side effects and tolerance, follow-up pregnancy and production, the
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Pain before and after surgery | 01/2005~12/2015
  Visual analogue scale ranges from 0 to 10 points, with higher scores indicative of more pain. We measure it before the surgery and follow it after intervention one month, three months and six months seperately.

SECONDARY OUTCOMES:
Hemoglobin | 01/2005~12/2015
  Preoperative serum hemoglobin levels were measured in women diagnosed by ultrasound or with endometriosis, adenomyosis, leiomyomas. We also follow up after intervention one month, three months and six months seperately.
  The normal value is range 12-15g/dl.
Tumor marker (CA-125) | 01/2005~12/2015
  Preoperative serum CA-125 levels were measured in women diagnosed by ultrasound or with endometriosis, adenomyosis, leiomyomas. We also follow up after intervention one month, three months and six months seperately. The normal value is less than 35 U/mL.
Ultrasound image tracking | 01/2005~12/2015
  Ovary endoemtriosis definition : Well-circumscribed thick-walled unilocular cyst that contains homogeneous low-level internal echoes ground glass. We measure it according to guideline Systematic approach to sonographic evaluation of the pelvis in women with suspected endometriosis, including terms,definitions and measurements: a consensus opinion from theInternational Deep Endometriosis Analysis (IDEA) group Adenomyosis definition : Asymmetrical myometrial thickening Globular shape, ill defined endometrial/ myometrial interface and linear striations. We measure it according to guideline Systematic approach to sonographic evaluation of the pelvisin women with suspected endometriosis, including terms,definitions and measurements: a consensus opinion from theInternational Deep Endometriosis Analysis (IDEA) group

CONTACTS AND LOCATIONS:
Overall Officials: Peng-Hui Wang, MD, PhD, Study Chair — pongpongwang@gmail.com
Locations (1):
- Peng-Hui Wang, Taipei County, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No